CLINICAL TRIAL: NCT05417295
Title: Position Related Bronchial Injury Caused by Bronchial Cuff of Double Lumen Endotracheal Tube
Brief Title: Bronchial Injury Caused by Bronchial Cuff
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KMUHIRB-F(II)-20210164
Record Dates: First submitted 2022-05-19; First posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-03

CONDITIONS: Bronchial Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inflating air into the bronchial cuff before changing position (Experimental): Before changing from supine position to lateral position, inflate air into the bronchial cuff of double lumen endotracheal tube (DLT) and adjust cuff pressure to 25-30 mmHg.
  Interventions: Procedure: Inflating air into the bronchial cuff before changing position
- Inflating air into the bronchial cuff after changing position (Placebo Comparator): Do not inflate air into the bronchial cuff before changing position.
  Interventions: Procedure: Inflating air into the bronchial cuff after changing position

INTERVENTIONS:
Procedure: Inflating air into the bronchial cuff before changing position — Inflating air into the bronchial cuff before or after changing position
  Arms: Inflating air into the bronchial cuff before changing position
Procedure: Inflating air into the bronchial cuff after changing position — Inflating air into the bronchial cuff after changing position
  Arms: Inflating air into the bronchial cuff after changing position

SUMMARY:
Double lumen endotracheal tubes (DLT) are wildly used to maintain independent lung ventilation during thoracic surgery. Our aim is to assess whether the DLT bronchial cuff inflated or not is associated with tube displacement and bronchial mucosal injury while changing position.

DETAILED DESCRIPTION:
Experiment group: Before changing from supine position to lateral position, inflate air into the bronchial cuff of double lumen endotracheal tube (DLT) and adjust cuff pressure to 25-30 mmHg.

Control group: Do not inflate air into the bronchial cuff before changing position.

Main result: Degree of left bronchial mucosal injury. Secondary result: Displacement of double lumen endotracheal tube after changing position.

All patients receive general anesthesia and are intubated with left DLT in the supine position. The fiberoptic bronchoscope is used to check the position via tracheal lumen of DLT. The bronchial lumen is placed at the left bronchus and the edge of bronchial cuff is visible by fiberscope.

Before changing position, the bronchial cuff of experiment group is inflated with air and adjusted cuff pressure to 25-30 mmHg. Both groups of patient's neck are fixed by neck collar in order to prevent displacement of DLT by neck rotation. After changing into lateral position, the assistant inflates 2 ml of into the bronchial cuff of control group and adjust cuff pressure to 25-30 mmHg. The investigator, blinded to the tube assignments, uses the fiberoptic bronchoscope to check position of the tube again via tracheal lumen of DLT and record the distance of displacement.

At the end of the surgery, both lumens of DLT are sucked and bronchial cuffs are deflated. After pulling out 3 cm of the DLT, the patient is changed into supine position and the fiberoptic bronchoscope is used to check the degree of bronchial injury.

ELIGIBILITY:
Inclusion Criteria:

* Patients receive elective thoracoscopic wedge resection in the lateral position and are intubated with left side double lumen endotracheal tube.

Exclusion Criteria:

* ASA status > III, coagulopathy, known airway damage, difficult intubation, tracheostomy, double lumen endotracheal tube is displaced during operation which interferes one lung ventilation and needs to be adjusted.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Left bronchial mucosal injury | Before extubation
  Degree of left bronchial mucosal injury is recorded via bronchoscope. Intact = 0 Redness = 1 Swelling = 2 hematoma = 3 Bleeding = 4

SECONDARY OUTCOMES:
Displacement of double lumen endotracheal tube | After changing into lateral position
  Displacement of double lumen endotracheal tube after changing position